CLINICAL TRIAL: NCT03427164
Title: Ultrasound Elastography Assessment of Spleen and Liver Stiffness Before and After Transjugular Intrahepatic Portosystemic Shunt (TIPS) Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004361
Record Dates: First submitted 2018-02-02; First posted 2018-02-09 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Portal Hypertension
Keywords: Transjugular Intrahepatic Portosystemic Shunt; TIPS; cirrhosis; hepatitis; portal vein thrombosis; Budd-Chiari Disease; Elastography
MeSH Terms: conditions — Hypertension, Portal; Fibrosis; Hepatitis | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TIPS (Experimental): Participants will have measurements taken of spleen stiffness before and after TIPS. Participation will last about 12 months, with visits at 1-2 weeks post-TIPS, 3 months, 6 months, and 12 months.
  Interventions: Procedure: Transjugular Intrahepatic Portosystemic Shunt

INTERVENTIONS:
Procedure: Transjugular Intrahepatic Portosystemic Shunt — The TIPS procedures creates an artificial shunt from the portal vein to the hepatic vein. TIPS allows blood from the congested portal circulation to bypass the fibrotic liver and directly enter the systemic circulation.
  Other Names: TIPS

SUMMARY:
The primary purpose of this project is to determine if acute monitoring of shunt patency via ultrasound elastography measurements of splenic stiffness before and after TIPS placement results in reduced morbidity and mortality from shunt failure.

DETAILED DESCRIPTION:
Portal hypertension is a condition that is caused by various disorders of the liver, including cirrhosis, hepatitis, portal vein thrombosis, or Budd-Chiari Disease. Portal hypertension can lead to the accumulation of fluid in the abdomen, called ascites, or put patients at risk for bleeding of the esophagus, stomach, and bowel. In certain patients, portal hypertension is treated by placement of a Transjugular Intrahepatic Portosystemic Shunt (TIPS).

Elastography is a newer exam which measures the consistency, or softness/stiffness, of various organs in the body. It is performed with ultrasound by sliding a transducer across the abdomen. Elastography is most commonly used to evaluate the liver, as disorders that cause damage to the liver result in stiffer liver tissue. The spleen has also been shown to get stiffer in the setting of portal hypertension.

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo TIPS placement at the University of Kansas Medical Center (KUMC) are eligible for participation in this study

Exclusion Criteria:

* Patients under 18 years of age
* Patients with prior splenectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Spleen stiffness | Change from Baseline to 2 weeks post-procedure
  The spleen stiffness will be measured before and after TIPS placement. Spleen stiffness is measured using US elastography and is reported in m/sec.

SECONDARY OUTCOMES:
Change in spleen stiffness | Change from Baseline to Month 12
  The spleen stiffness will be measured before and after TIPS placement. Spleen stiffness is measured using US elastography and is reported in m/sec.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Jones, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No